CLINICAL TRIAL: NCT00823888
Title: Mechanics of Knee Bracing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The New England Baptist Hospital (Other)
Collaborators: Boston University (Other); Spaulding Rehabilitation Hospital (Other)
Responsible Party: William F Harvey, MD, New England Baptist Hospital
Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NEBH 2008-012
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Osteoarthritis, Knee
Keywords: Knee Osteoarthritis; pneumatic bracing
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: pneumatic brace — pneumatic knee brace with three trial conditions: air bladders inflated at 0psi, 7 psi, and 12 psi

SUMMARY:
The overall objective of this project is to determine whether the provision of a pneumatic knee brace in patients with medial knee osteoarthritis (OA) improves knee mechanics. Secondary objectives will be to assess if the brace relieves knee pain and improves function. We will test the hypothesis that compared to the control treatment (see below for the definition) the use of a pneumatic knee brace is effective in medial knee OA.

DETAILED DESCRIPTION:
This study is closed to enrollment and in the data analysis phase

ELIGIBILITY:
Inclusion Criteria:

* knee pain, aching or stiffness on most of the past 30 days
* x-ray verified predominant medial tibiofemoral osteoarthritis (TFOA)
* overall pain that is due to the medial TFOA (versus being referred from the back, hips, or other pre-existing conditions)
* ambulatory persons

Exclusion Criteria:

* use of a crutch, walker, or wheelchair or cane more than 50% of the time
* history of Deep Vein Thrombosis
* Pain emanating more from back or hip than from knee
* Low pain score on WOMAC
* predominant patellofemoral disease or knee pathology other than medial compartment OA likely to be causing their knee pain.
* Planning to move from area within 1 month of study screening.
* Unable to fit the brace properly
* BMI greater than 35
* corticosteriod injections in the past month
* Bilateral total knee replacements or plan for TKR
* Other types of arthritis including Rheumatoid Arthritis, Systemic Lupus Erythematosus, gout, psoriatic arthritis, pseudogout.
* woman who are pregnant (due to x-rays taken to determine eligibility)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To undertake a clinical trial in patients with medial knee OA to determine whether provision of a pneumatic knee brace leads to a reduced adduction moment during the time of this treatment than during the use of a control treatment. | At study visit

SECONDARY OUTCOMES:
To undertake a clinical trial in patients with medial knee OA to determine whether provision of a pneumatic knee brace leads to a lower pain score and improved function during the time of this treatment than during the use of a control treatment. | During study visit

CONTACTS AND LOCATIONS:
Overall Officials: William F Harvey, MD, Principal Investigator — New England Baptist Hospital, Tufts Medical Center
Locations (1):
- New England Baptist Hospital, Boston, Massachusetts, United States